CLINICAL TRIAL: NCT02909153
Title: Single Ascending Dose Study of Intraperitoneal Triferic (Ferric Pyrophosphate Citrate) in Patients on Chronic Peritoneal Dialysis
Brief Title: Study of Intraperitoneal Triferic in Patients on Chronic Peritoneal Dialysis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rockwell Medical Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RMFPC-17
Record Dates: First submitted 2016-09-19; First posted 2016-09-21 (Estimated); Results first posted 2019-08-08 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Peritoneal Dialysis (PD); Anemia; Chronic Kidney Disease
Keywords: Triferic; ferric pyrophosphate citrate (FPC); peritoneal dialysis; anemia; chronic kidney disease
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic | interventions — ferric pyrophosphate; spleen fibrinolytic proteinase (human)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- single dose of Triferic in the peritoneal dialysis solution (Experimental): The patient will receive a single dose of Triferic in the peritoneal dialysis solution (IP) during a long (12 hour) peritoneal dialysis dwell. Each Cohort will receive a different ascending IP dose ( 5 mg/L, 12.5 mg/L, 20 mg/L). Blood samples will be drawn periodically over a 12 hour period for analysis.
  Interventions: Drug: Triferic
- single IV dose of Triferic 6.6 mg over a 4 hour period (Experimental): The patient will receive a single 6.6 mg intravenous (IV) dose of Triferic in the over a 4 hour period. All Cohorts will receive the same IV dose. Blood samples will be drawn periodically over a 12 hour period for analysis.
  Interventions: Drug: Triferic

INTERVENTIONS:
Drug: Triferic — Triferic is an iron salt that is approved by the FDA for the maintenance of hemoglobin in patients with end stage kidney disease on hemodialysis. It is experimental in this study because it has not yet been approved for patients on chronic peritoneal dialysis.
  Other Names: ferric pyrophosphate citrate; FPC

SUMMARY:
The main purpose is to determine the pharmacokinetic (PK) profile, maximum concentration (Cmax) and Area Under the Concentration Time Curve (AUC0-t) of Triferic iron administered intraperitoneally in patients with chronic kidney disease on peritoneal dialysis (CKD-5 PD). It is an open label, dose escalation study.

DETAILED DESCRIPTION:
This is a phase 1, open-label, dose escalation study assessing the pharmacokinetic (PK) profile, maximum concentration (Cmax) and Area Under the Concentration Time Curve (AUC0-t) of Triferic iron administered intraperitoneally in chronic kidney disease patients on peritoneal dialysis (Continuous Cycling Peritoneal Dialysis (CCPD) or Continuous Ambulatory Peritoneal Dialysis (CAPD)).

Screening can be up to 4 weeks, and the enrollment period is approximately one week. There are two treatment (dosing) visits and one follow-up visit during the enrollment period.

At each treatment visit, the patients will be randomly assigned to receive either a single ascending dose of Triferic administered intraperitoneal (IP) during a long (12 hour) peritoneal dialysis dwell or a single 6.6 mg dose of Triferic administered IV over 4 hours. Blood samples will be obtained at defined times over 12 hours to establish the total serum iron PK of IP Triferic as well as the clinical serum iron profile.

The IP dose of the first Cohort will be 5 mg Triferic iron/liter IP. Subsequent Cohort IP doses will be 12.5 mg Triferic iron/liter, and 20 mg Triferic iron/liter, with the final Cohort dose to be determined (TBD). The IV dose will be 6.6. mg for all Cohorts. Six patients will be enrolled in each Cohort, with enrollment in the subsequent (higher dose) Cohort not being initiated until the completion and evaluation of the previous (lower dose) Cohort.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be able to provide informed consent and have personally signed and dated the study written informed consent document before completing any study-related procedures.
2. The patient must be 18-75 years of age inclusive at the time of consent.
3. Have a diagnosis of End Stage Renal Disease and have been on Peritoneal Dialysis for at least 3 months (CAPD or CCPD) prior to Screening.
4. Be in a stable clinical condition during the four weeks immediately prior to Screening Period as demonstrated by medical history, physical examination and laboratory testing
5. Have a blood hemoglobin concentration above 9.5 g/dL.
6. Have a total iron binding capacity (TIBC) of ≥ 175 µg/dL.
7. Have not experienced peritonitis episodes in the last 3 months prior to Screening.
8. The patient must agree to discontinue all iron preparations for 14 days prior to Study PD #1/Day 1.
9. Female patients must be nonpregnant and not breastfeeding. They must either have been amenorrheic for the past year or agree to not become pregnant by continuous use of an effective birth control method acceptable to the Investigator for the duration of their participation in the study.

Exclusion Criteria:

1. The patient has had an red blood cell (RBC) or whole blood transfusion within 4 weeks prior to Screening.
2. The patient has had administration of IV or oral iron supplements (including multivitamins with iron) within 14 days prior to Study PD #1/Day 1.
3. The patient has known active bleeding from any site (e.g., gastrointestinal, hemorrhoid, nasal, pulmonary, etc.).
4. The patient has a living kidney donor identified or living-donor kidney transplant scheduled to occur during study participation. (Note: Patients awaiting deceased-donor transplant need not be excluded.)
5. The patient is scheduled to have a surgical procedure during the study.
6. The patient has had a hospitalization within the 4 weeks prior to Screening (except for vascular access surgery) that, in the opinion of the Investigator, confers a significant risk of hospitalization during the course of the study.
7. The patient has a history of noncompliance with the dialysis regimen in the opinion of the Investigator.
8. The patient has a known ongoing inflammatory disorder (other than chronic kidney disease), such as systemic lupus erythematosus, rheumatoid arthritis, or other collagen-vascular disease, that currently requires systemic anti-inflammatory or immunomodulatory therapy.
9. The patient has any current febrile illness (e.g., oral temperature ≥100.4°F, 38.0°C). (Patients may subsequently become eligible at least 1 week after resolution of the illness.)
10. The patient has known bacterial, tuberculosis, fungal, viral, or parasitic infection requiring anti-microbial therapy or anticipated to require anti-microbial therapy during the patient's participation in this study.
11. The patient is known to be positive for HIV, hepatitis B, or hepatitis C (viral testing is not required as part of this protocol).
12. The patient has cirrhosis of the liver based on histological criteria or clinical criteria (e.g., presence of ascites, esophageal varices, multiple spider nevi, or history of hepatic encephalopathy).
13. The patient has alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) levels consistently greater than twice the upper limit of normal at any time during the two months prior to Study PD #1/Day 1.
14. The patient currently has any malignancy other than basal or squamous cell skin cancer.
15. The patient has a history of drug or alcohol abuse within the 6 months prior to Screening.
16. The patient participated in an investigational drug study within 30 days prior to Study PD #1/Day 1.
17. The patient has any condition that, in the opinion of the Investigator, would make it unlikely for the patient to complete the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-01; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond D Pratt, MD, FACP, Study Director — Rockwell Medical, Inc

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Patients in Cohort 1 received 2 doses of Triferic in a randomized, cross-over design. The doses were Triferic 5 mg Fe/L in Dianeal PD solution and Triferic 6.6 mg Fe via 4-hour IV infusion, with 48 hours separating the start of each dose.
- Cohort 2: Patients in Cohort 2 received 2 doses of Triferic in a randomized, cross-over design. The doses were Triferic 12.5 mg Fe/L in Dianeal PD solution and Triferic 6.6 mg Fe via 4-hour IV infusion, with 48 hours separating the start of each dose.
- Cohort 3: Patients in Cohort 3 received 2 doses of Triferic in a randomized, cross-over design. The doses were Triferic7. 5 mg Fe/L in Dianeal PD solution and Triferic 6.6 mg Fe via 4-hour IV infusion, with 48 hours separating the start of each dose.
- Cohort 4: Patients in Cohort 4 received 2 doses of Triferic in a randomized, cross-over design. The doses were Triferic 5 mg Fe/L in Extraneal PD solution and Triferic 6.6 mg Fe via 4-hour IV infusion, with 48 hours separating the start of each dose.
- Cohort 5: Patients in Cohort 5 received 2 doses of Triferic in a randomized, cross-over design. The doses were Triferic 2.5 mg Fe/L in Extraneal PD solution and Triferic 6.6 mg Fe via 4-hour IV infusion, with 48 hours separating the start of each dose.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Started | 6 | 6 | 6 | 6 | 6
Triferic in Dianeal PD Solution (Cohort 1: 5 mg Fe/L Triferic, Cohort 2: 12.5 mg Fe/L Triferic, Cohort 3: 7.5 mg Fe/L Triferic) | 6 | 6 | 6 | 0 | 0
Triferic 6.6mg Fe Via 4hr IV Infusions | 6 | 5 | 6 | 6 | 6
Triferic in Extraneal PD Solution (Cohort 4: dosed Triferic 5 mg Fe/L, Cohort 5: dosed Triferic 2.5 mg Fe/L) | 0 | 0 | 0 | 6 | 6
Completed | 6 | 5 | 6 | 6 | 6
Not Completed | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (8.2) | 45.8 (19.6) | 56.7 (10.2) | 45.2 (21.5) | 56.3 (15.9) | 53.3 (16.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 4 | 2 | 3 | 14
  Male | 5 | 2 | 2 | 4 | 3 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 3 | 3 | 3 | 14
  Not Hispanic or Latino | 3 | 4 | 3 | 3 | 3 | 16
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 1 | 2 | 5
  White | 6 | 4 | 6 | 4 | 4 | 24
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 6 | 6 | 6 | 30

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK) of Triferic Iron Administered in Patients on Chronic Peritoneal Dialysis: Maximum Concentration (Cmax) of Serum Total Iron After Intraperitoneal Administration of Triferic
Description: The PK will be done by assessing the mean absolute Cmax of Triferic iron administered intraperitoneally in patients with chronic kidney disease on peritoneal dialysis (CKD-5 PD).
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 12 hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per deciliter
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
microgram per deciliter | 164 (25.0) | 213 (3.78) | 153 (32.1) | 163 (19.4) | 105 (15.9)

2. Primary Outcome: Pharmacokinetics (PK) of Triferic Iron Administered in Patients on Chronic Peritoneal Dialysis: Area Under the Concentration Curve (AUC) Last of Serum Total Iron After Intraperitoneal Administration of Triferic
Description: The PK will be done by assessing the AUC from time zero to the time of the last quantified concentration (AUClast) of Triferic iron administered intraperitoneally in patients with chronic kidney disease on peritoneal dialysis (CKD-5 PD).
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 12 hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours x micrograms/ deciliters
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6
hours x micrograms/ deciliters | 1690 (27.9) | 2220 (9.84) | 2560 (33.0) | 2510 (41.8) | 2260 (23.9)

3. Primary Outcome: Pharmacokinetics (PK) of Triferic Iron Administered in Patients on Chronic Peritoneal Dialysis: Area Under the Concentration Curve (AUC) 0 - 12 of Serum Total Iron After Intraperitoneal Administration of Triferic
Description: The PK will be done by assessing the AUC from time zero to 12 hours after infusion (AUC0-12) of Triferic iron administered intraperitoneally in patients with chronic kidney disease on peritoneal dialysis (CKD-5 PD).
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 12 hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours x micrograms/ deciliters
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6
hours x micrograms/ deciliters | 1690 (27.9) | 2220 (9.84) | 1580 (41.8) | 1610 (32.3) | 1050 (20.9)

4. Primary Outcome: Pharmacokinetics (PK) of Triferic Iron Administered in Patients on Chronic Peritoneal Dialysis: Maximum Concentration (Cmax) of Serum Total Iron After Intravenous Administration of Triferic
Description: The PK will be done by assessing the mean absolute Cmax of Triferic iron administered intravenously in patients with chronic kidney disease on peritoneal dialysis (CKD-5 PD).
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 12 hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/ deciliters
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6
micrograms/ deciliters | 217 (41.9) | 203 (32.6) | 183 (30.3) | 254212 (14.7) | 177 (30.8)

5. Primary Outcome: Pharmacokinetics (PK) of Triferic Iron Administered in Patients on Chronic Peritoneal Dialysis: Area Under the Concentration Curve (AUC) Last of Serum Total Iron After Intravenous Administration of Triferic
Description: The PK will be done by assessing the AUC from time zero to the time of the last quantified concentration (AUClast) of Triferic iron administered intravenously in patients with chronic kidney disease on peritoneal dialysis (CKD-5 PD).
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 12 hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours* micrograms/ deciliters
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6
hours* micrograms/ deciliters | 1750 (33.8) | 1730 (28.2) | 2160 (30.0) | 3060 (33.6) | 2840 (35.7)

6. Primary Outcome: Pharmacokinetics (PK) of Triferic Iron Administered in Patients on Chronic Peritoneal Dialysis: Area Under the Concentration Curve (AUC) 0-12 of Serum Total Iron After Intravenous Administration of Triferic
Description: The PK will be done by assessing the AUC from time zero to 12 hours after the infusion (AUC0-12) of Triferic iron administered intravenously in patients with chronic kidney disease on peritoneal dialysis (CKD-5 PD).
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 12 hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours* micrograms/ deciliters
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6
hours* micrograms/ deciliters | 1750 (33.8) | 1730 (28.2) | 1530 (41.3) | 1890 (20.9) | 1560 (31.7)

7. Secondary Outcome: Bioavailability of Triferic Iron Administered Via PD Solution: F(Cmax)
Description: The bioavailability (F) of the maximum serum iron concentration (Cmax) of Triferic iron was quantified for the peritoneal dialysis dose of Triferic for all cohorts.
Time Frame: 12 hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percent of bioavailability
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6
percent of bioavailability | 47.7 (28.3) | 26.5 (30.9) | 34.9 (25.2) | 62.6 (17.3) | 74.6 (25.9)

ADVERSE EVENTS:
Time Frame: Adverse events data was collected from the date of enrollment through the completion of the follow-up study visit. This timeframe was approximately 5 days.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 1/6 | 2/6 | 1/6 | 1/6 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=6) | Cohort 2 (N=6) | Cohort 3 (N=6) | Cohort 4 (N=6) | Cohort 5 (N=6)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Groin Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2016-11-21): https://cdn.clinicaltrials.gov/large-docs/53/NCT02909153/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-26): https://cdn.clinicaltrials.gov/large-docs/53/NCT02909153/SAP_001.pdf